CLINICAL TRIAL: NCT02395042
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study, Evaluating Safety and Efficacy of LiRIS® 400 mg in Females With Interstitial Cystitis With Hunner's Lesions
Brief Title: A Safety and Efficacy Study of LiRIS® in Females With Interstitial Cystitis With Hunner's Lesions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201025-001
Record Dates: First submitted 2015-03-17; First posted 2015-03-20 (Estimated); Results first posted 2018-10-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-08

CONDITIONS: Cystitis, Interstitial; Ulcer
MeSH Terms: conditions — Cystitis, Interstitial; Ulcer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- LiRIS Placebo, LiRIS Placebo (Tx 1)/LiRIS® (Tx 2) (Placebo Comparator): Treatment 1 Period (Tx 1): Matching placebo device to the LiRIS inserted into the bladder by cystoscopy on Day 10 and then removed and a second matching placebo device to the LiRIS inserted into the bladder by cystoscopy on Day 14 and removed on Day 28. Treatment 2 Period (Tx 2): optional LiRIS® (continuous release of lidocaine) 400 mg inserted into the bladder by cystoscopy on Day 0 and removed on Day 14.
  Interventions: Drug: LiRIS®
- LiRIS®, LiRIS® (Tx 1)/LiRIS® (Tx 2) (Experimental): Treatment 1 Period: LiRIS® (continuous release of lidocaine) 400 mg inserted into the bladder by cystoscopy on Day 0 then removed and a second LiRIS® 400 mg inserted into the bladder on Day 14 and removed on Day 28. Treatment 2 Period: optional LiRIS® (continuous release of lidocaine) 400 mg inserted into the bladder by cystoscopy on Day 0 and then removed on Day 14.
  Interventions: Drug: LiRIS®; Drug: LiRIS Placebo
- LiRIS Placebo, LiRIS® (Tx 1)/ LiRIS® (Tx 2) (Experimental): Treatment 1 Period: Matching placebo device to the LiRIS inserted into the bladder by cystoscopy on Day 0 and then removed and LiRIS® (continuous release of lidocaine) 400 mg inserted into the bladder by cystoscopy on Day 14 then removed on Day 28. Treatment 2 Period: optional LiRIS® 400 mg inserted into the bladder by cystoscopy on Day 0 then removed on Day 14.
  Interventions: Drug: LiRIS®; Drug: LiRIS Placebo

INTERVENTIONS:
Drug: LiRIS® — LiRIS® is a drug-device combination product which is placed in the bladder during cystoscopy and remains in the bladder, gradually releasing lidocaine until removed from the bladder via cystoscopy.
Drug: LiRIS Placebo — LiRIS placebo is a drug-device combination product, matching the LiRIS® which is placed in the bladder during cystoscopy, remains in the bladder until removed from the bladder via cystoscopy
  Arms: LiRIS Placebo, LiRIS® (Tx 1)/ LiRIS® (Tx 2); LiRIS®, LiRIS® (Tx 1)/LiRIS® (Tx 2)

SUMMARY:
This is a safety and efficacy study of LiRIS® in females with interstitial cystitis with Hunner's lesions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of interstitial cystitis with Hunner's lesions/ulcers

Exclusion Criteria:

* Previous treatment with LiRIS®
* Interstitial cystitis/bladder pain syndrome, without Hunner's lesions/ulcers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-04-15 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2017-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Till Geib, Study Director — Allergan
Locations (19):
- United States (17):
  - Tri Valley Urology Medical Group, Murrieta, California
  - Sutter Institute for Medical Research, Vacaville, California
  - Women's Health Specialty Care, Farmington, Connecticut
  - Atlanta Medical Research Institute, Alpharetta, Georgia
  - Anne Arundel Urology, P.A., Annapolis, Maryland
  - Chesapeake Urology Research Associates, Baltimore, Maryland
  - Beyer Research, Kalamazoo, Michigan
  - Beaumont Health System, Royal Oak, Michigan
  - Washington University School of Medicine Department of Surgery, St Louis, Missouri
  - Western New York Urology Associates, LLC, Cheektowaga, New York
  - McKay Urology, Charlotte, North Carolina
  - Eastern Urological Associates, PA, Greenville, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - MetroHealth System/Center for Advanced Gynecology, Cleveland, Ohio
  - Philadelphia Urosurgical Associates, Philadelphia, Pennsylvania
  - University of Washington, Seattle, Washington
  - Aurora Health Care, West Allis, Wisconsin
- Canada (2):
  - Silverado Research Inc, Victoria, British Columbia
  - Sunnybrook Health Science Centre, Toronto, Ontario

REFERENCES:
- [Derived] Evans R, Kohan A, Moldwin R, Radecki D, Geib T, Peters KM. Safety, tolerability, and efficacy of LiRIS 400 mg in women with interstitial cystitis/bladder pain syndrome with or without Hunner lesions. Neurourol Urodyn. 2021 Sep;40(7):1730-1739. doi: 10.1002/nau.24702. Epub 2021 Jul 20. PMID 34288094

RESULTS

PARTICIPANT FLOW:
Groups:
- LiRIS Placebo, LiRIS Placebo (Tx 1)/LiRIS® (Tx 2): Treatment 1 Period: Matching placebo device to the LiRIS inserted into the bladder by cystoscopy on Day 10 and then removed and a second matching placebo device to the LiRIS inserted into the bladder by cystoscopy on Day 14 and removed on Day 28. Treatment 2 Period: optional LiRIS® (continuous release of lidocaine) 400 mg inserted into the bladder by cystoscopy on Day 0 and removed on Day 14.
Period: Treatment 1 Period
Arm/Group | LiRIS Placebo, LiRIS Placebo (Tx 1)/LiRIS® (Tx 2) | LiRIS®, LiRIS® (Tx 1)/LiRIS® (Tx 2) | LiRIS Placebo, LiRIS® (Tx 1)/ LiRIS® (Tx 2)
Started | 12 | 31 | 16
Completed | 9 | 25 | 14
Not Completed | 3 | 6 | 2
Not completed — Adverse Event | 1 | 3 | 1
Not completed — Lack of Efficacy | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Other Miscellaneous Reasons | 0 | 2 | 1
Period: Treatment 2 Period
Arm/Group | LiRIS Placebo, LiRIS Placebo (Tx 1)/LiRIS® (Tx 2) | LiRIS®, LiRIS® (Tx 1)/LiRIS® (Tx 2) | LiRIS Placebo, LiRIS® (Tx 1)/ LiRIS® (Tx 2)
Started | 10 (Not all participants participated in Treatment 2 Period.) | 24 (Not all participants participated in Treatment 2 Period.) | 13 (Not all participants participated in Treatment 2 Period.)
Completed | 9 | 23 | 13
Not Completed | 1 | 1 | 0
Not completed — Lack of Efficacy | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-treat (mITT) Population included all randomized participants who had the investigational product inserted.
Groups:
- Total: Total of all reporting groups
Arm/Group | LiRIS Placebo, LiRIS Placebo (Tx 1)/LiRIS® (Tx 2) | LiRIS®, LiRIS® (Tx 1)/LiRIS® (Tx 2) | LiRIS Placebo, LiRIS® (Tx 1)/ LiRIS® (Tx 2) | Total
Number analyzed (Participants) | 12 | 31 | 16 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.58 (12.09) | 57.65 (12.76) | 57.31 (14.25) | 56.73 (12.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 31 | 16 | 59
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 8 | 29 | 16 | 53
  Black | 3 | 1 | 0 | 4
  Asian | 0 | 1 | 0 | 1
  Hispanic | 1 | 0 | 0 | 1
Daily Average Bladder Pain Numeric Rating Scale (NRS) [Mean (Full Range); unit: score on a scale] — The participant recorded their daily bladder pain score over the previous 24-hour period on a 7-day pain assessment tool as measured by an NRS on an 11-point scale where 0=no pain to 10=worst pain imaginable. The daily pain scores over the 7-day period were averaged. Population: Modified Intent-to-Treat population, all participants who were randomized and received Treatment 1, with available baseline data.
  score on a scale
    number analyzed (Participants) | 11 | 28 | 14 | 53
    (all) | 6.0 [4.3 to 8.0] | 5.5 [3.2 to 9.3] | 5.6 [4.1 to 7.8] | 5.7 [3.2 to 9.3]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Daily Average Bladder Pain Numeric Rating Scale (NRS)
Description: The participant recorded their daily bladder pain score over the previous 24-hour period on a 7-day pain assessment tool as measured by an NRS on an 11-point scale where 0=no pain to 10=worst pain imaginable. The daily pain scores over the 7-day period were averaged. A negative change from Baseline indicates improvement. An analysis of covariance (ANCOVA) model with Baseline value as a covariate and treatment group and stratification (baseline bladder pain NRS: ≤ 5 or > 5) as factors was used for analysis.
Time Frame: Baseline (Day -7 to Day 0) to Week 4
Population: Modified Intent-to-Treat population, all participants who were randomized and received Treatment 1, with data available for analysis.
Measure: Least Squares Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | LiRIS Placebo, LiRIS Placebo (Tx 1)/LiRIS® (Tx 2) | LiRIS®, LiRIS® (Tx 1)/LiRIS® (Tx 2) | LiRIS Placebo, LiRIS® (Tx 1)/ LiRIS® (Tx 2)
Number analyzed (Participants) | 9 | 26 | 10
score on a scale | -1.6 [-2.68 to -0.45] | -2.7 [-3.36 to -2.06] | -2.5 [-3.53 to -1.44]
Statistical Analysis 1: Comparison: LiRIS Placebo, LiRIS Placebo (Tx 1)/LiRIS® (Tx 2) vs LiRIS®, LiRIS® (Tx 1)/LiRIS® (Tx 2); Test type: Superiority; p = 0.142, ANCOVA; ANCOVA model with baseline value as a covariate and treatment group and stratification (baseline bladder pain NRS: ≤ 5 or > 5) as factors; Least Squares Mean Difference = -1.15
Statistical Analysis 2: Comparison: LiRIS Placebo, LiRIS Placebo (Tx 1)/LiRIS® (Tx 2) vs LiRIS Placebo, LiRIS® (Tx 1)/ LiRIS® (Tx 2); Test type: Superiority; p = 0.319, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.92

2. Secondary Outcome: Change From Baseline in the Number of Hunner's Lesions
Description: During each cystoscopy, the investigator counted the number of lesions visible while performing the bladder scan. A negative change from Baseline indicates improvement (less lesions). An ANCOVA model with Baseline value as a covariate and treatment group and stratification (baseline bladder pain NRS: ≤ 5 or > 5) as factors was used for analysis.
Time Frame: Baseline (Day 0) to Week 4
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Hunner's lesions
Arm/Group | LiRIS Placebo, LiRIS Placebo (Tx 1)/LiRIS® (Tx 2) | LiRIS®, LiRIS® (Tx 1)/LiRIS® (Tx 2) | LiRIS Placebo, LiRIS® (Tx 1)/ LiRIS® (Tx 2)
Number analyzed (Participants) | 8 | 18 | 12
Hunner's lesions | 0.8 [-0.04 to 1.7] | -0.6 [-1.21 to -0.05] | -0.2 [-0.87 to 0.50]
Statistical Analysis 1: Comparison: LiRIS Placebo, LiRIS Placebo (Tx 1)/LiRIS® (Tx 2) vs LiRIS®, LiRIS® (Tx 1)/LiRIS® (Tx 2); Test type: Superiority; p = 0.024, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -1.46
Statistical Analysis 2: Comparison: LiRIS Placebo, LiRIS Placebo (Tx 1)/LiRIS® (Tx 2) vs LiRIS Placebo, LiRIS® (Tx 1)/ LiRIS® (Tx 2); Test type: Superiority; p = 0.137, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -1.02

3. Secondary Outcome: Change From Baseline in Composite Score of Hunner's Lesions Calculated Based on Number, Size, and Severity of Lesions
Description: A standardized video capture protocol for bladder mapping was followed to assess any changes in the number, the size and the severity, of lesions during the study as a result of treatment. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Week 4
Population: Data for the planned composite Hunner's Lesions score were supposed to be generated based on digital images by a software algorithm, but the system never worked and no data were generated.
Arm/Group | LiRIS Placebo, LiRIS Placebo (Tx 1)/LiRIS® (Tx 2) | LiRIS®, LiRIS® (Tx 1)/LiRIS® (Tx 2) | LiRIS Placebo, LiRIS® (Tx 1)/ LiRIS® (Tx 2)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment 1 Period Up to Week 20 and Treatment 2 Period Up to 52 days
Description: Due to study design the Non-serious Adverse Event (AE) tables are reported separately for Treatment 1 Period and Treatment 2 Period. A result of 0 in an arm means that there were no participants in that arm at a threshold of >=5% for the preferred term.
Groups:
- LiRIS Placebo, LiRIS Placebo (Tx 1): Treatment 1 Period: Matching placebo device to the LiRIS inserted into the bladder by cystoscopy on Day 10 and then removed and a second matching placebo device to the LiRIS inserted into the bladder by cystoscopy on Day 14 and removed on Day 28. Adverse events (AEs) reported in Tx 1.
- LiRIS®, LiRIS® (Tx 1): Treatment 1 Period: LiRIS® (continuous release of lidocaine) 400 mg inserted into the bladder by cystoscopy on Day 0 then removed and a second LiRIS® 400 mg inserted into the bladder on Day 14 and removed on Day 28. AEs reported in Tx 1.
- LiRIS Placebo, LiRIS® (Tx 1): Treatment 1 Period: Matching placebo device to the LiRIS inserted into the bladder by cystoscopy on Day 0 and then removed and LiRIS® (continuous release of lidocaine) 400 mg inserted into the bladder by cystoscopy on Day 14 then removed on Day 28. AEs reported in Tx 1.
- LiRIS Placebo, LiRIS Placebo/LiRIS® (Tx 2): Treatment 1 Period: Matching placebo device to the LiRIS inserted into the bladder by cystoscopy on Day 10 and then removed and a second matching placebo device to the LiRIS inserted into the bladder by cystoscopy on Day 14 and removed on Day 28. Treatment 2 Period: optional LiRIS® (continuous release of lidocaine) 400 mg inserted into the bladder by cystoscopy on Day 0 and removed on Day 14. AEs reported in Tx 2.
- LiRIS®, LiRIS® /LiRIS® (Tx 2): Treatment 1 Period: LiRIS® (continuous release of lidocaine) 400 mg inserted into the bladder by cystoscopy on Day 0 then removed and a second LiRIS® 400 mg inserted into the bladder on Day 14 and removed on Day 28. Treatment 2 Period: optional LiRIS® (continuous release of lidocaine) 400 mg inserted into the bladder by cystoscopy on Day 0 and then removed on Day 14. AEs reported in Tx 2.
- LiRIS Placebo, LiRIS /LiRIS® (Tx 2): Treatment 1 Period: Matching placebo device to the LiRIS inserted into the bladder by cystoscopy on Day 0 and then removed and LiRIS® (continuous release of lidocaine) 400 mg inserted into the bladder by cystoscopy on Day 14 then removed on Day 28. Treatment 2 Period: optional LiRIS® 400 mg inserted into the bladder by cystoscopy on Day 0 then removed on Day 14. AEs reported in Tx 2.
Arm/Group | LiRIS Placebo, LiRIS Placebo (Tx 1) | LiRIS®, LiRIS® (Tx 1) | LiRIS Placebo, LiRIS® (Tx 1) | LiRIS Placebo, LiRIS Placebo/LiRIS® (Tx 2) | LiRIS®, LiRIS® /LiRIS® (Tx 2) | LiRIS Placebo, LiRIS /LiRIS® (Tx 2)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/31 | 0/16 | 0/10 | 0/24 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/31 | 0/16 | 0/10 | 0/24 | 0/13
Other Adverse Events (participants affected / at risk) | 9/12 | 21/31 | 10/16 | 4/10 | 2/24 | 3/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LiRIS Placebo, LiRIS Placebo (Tx 1) (N=12) | LiRIS®, LiRIS® (Tx 1) (N=31) | LiRIS Placebo, LiRIS® (Tx 1) (N=16) | LiRIS Placebo, LiRIS Placebo/LiRIS® (Tx 2) (N=10) | LiRIS®, LiRIS® /LiRIS® (Tx 2) (N=24) | LiRIS Placebo, LiRIS /LiRIS® (Tx 2) (N=13)
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LiRIS Placebo, LiRIS Placebo (Tx 1) (N=12) | LiRIS®, LiRIS® (Tx 1) (N=31) | LiRIS Placebo, LiRIS® (Tx 1) (N=16) | LiRIS Placebo, LiRIS Placebo/LiRIS® (Tx 2) (N=10) | LiRIS®, LiRIS® /LiRIS® (Tx 2) (N=24) | LiRIS Placebo, LiRIS /LiRIS® (Tx 2) (N=13)
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Medical device pain (General disorders) | 0 | 2 | 1 | 0 | 0 | 0
Suprapubic pain (General disorders) | 1 | 2 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 0 | 0 | 0
Medical device discomfort (General disorders) | 0 | 2 | 0 | 0 | 0 | 0
Thirst (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 5 | 2 | 0 | 0 | 1
Genital herpes (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 5 | 6 | 3 | 0 | 0 | 0
Bladder pain (Renal and urinary disorders) | 1 | 3 | 3 | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 4 | 2 | 0 | 0 | 0
Bladder discomfort (Renal and urinary disorders) | 0 | 4 | 0 | 0 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0
Urethral pain (Renal and urinary disorders) | 0 | 0 | 2 | 1 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urge incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Genital infection fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2016-04-28): https://cdn.clinicaltrials.gov/large-docs/42/NCT02395042/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-27): https://cdn.clinicaltrials.gov/large-docs/42/NCT02395042/SAP_001.pdf